CLINICAL TRIAL: NCT03204461
Title: Associatons of PCOS Phenotypes With Ectopic Lipids, Adipocytokines and Parameters of Insulin Resistance
Brief Title: Glucose Metabolism in Different PCOS Phenotypes
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Univ.Prof.Dr., Medical University of Vienna
Other Study IDs: PCOS-1090
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Polycystic Ovary Syndrome; Glucose Intolerance; Liver Fat; Glucose Metabolism Disorders
MeSH Terms: conditions — Polycystic Ovary Syndrome; Glucose Intolerance; Fatty Liver; Glucose Metabolism Disorders | interventions — Glucose Tolerance Test; Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCOS-NIH
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Other: 1H-magnetic resonance spectroscopy
- PCOS-Rotterdam
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Other: 1H-magnetic resonance spectroscopy
- Controls
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Other: 1H-magnetic resonance spectroscopy

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test (OGTT) — For the assessment of glucose metabolism, including beta-cell function and insulin sensitivity an 75g-OGTT was conducted.
Other: 1H-magnetic resonance spectroscopy — The amount of ectopic lipids in the liver, heart and the skeletal muscle was measured using 1H-magnetic resonance spectroscopy.

SUMMARY:
In the present study glucose metabolism and ectopic lipids in the liver, heart and muscle were investigated in women with the polycystic ovary syndrome (PCOS) and in healthy control subjects.

DETAILED DESCRIPTION:
In detail an oral glucose tolerance test (OGTT) was conducted in women with the PCOS defined by the Rotterdam and the NIH-criteria, as well as in healthy control subjects. In addition 1H-magnetic resonance spectroscopy and Imaging was used for the assessment of the ectopic lipid content in the liver, heart and skeletal muscle. The aim of the present study was to compare the glucose metabolism and the ectopic lipid conent in the liver, heart and muscle between women with the PCOS defined by the NIH-criteria, Rotterdam-criteria and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Women with the polycystic ovary Syndrome defined according to the Rotterdam and the NIH-criteria
* healthy control subjects

Exclusion Criteria:

* BMI>=40kg/m²
* Diagnosis of Diabetes in the PCOS-Group
* Diagnosis of Prediabetes or Diabetes in the control group

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the present study women with the Polycystic Ovary Syndrome, defined according to the NIH-criteria and the Rotterdam criteria were included. The control Group consisted of healthy volunteers without a diagnosis of prediabetes, Diabetes or the PCOS.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison of glucose metabolism between PCOS women and healthy control subjects, using data of the OGTT. | Up to 4 weeks
  In the present study the Glucose metabolism in PCOS women and control subjects was assessed with an OGTT. Therefore the dynamic levels of glucose, insulin and C-peptide were assessed during an extended OGTT for the calculation of Insulin resistance and beta-cell function. In addition an 1H-magnetic resonance spectroscopy was done for the assessment of the ectopic lipid content in the liver, heart and the skeletal muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Univ.Prof.Dr., Principal Investigator — Department of Internal Medicine III, Clinical Division of Endocrinology and Metabolism, Unit of Gender Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Leutner M, Gobl C, Wolf P, Maruszczak K, Bozkurt L, Steinbrecher H, Just-Kukurova I, Ott J, Egarter C, Trattnig S, Kautzky-Willer A. Pericardial Fat Relates to Disturbances of Glucose Metabolism in Women with the Polycystic Ovary Syndrome, but Not in Healthy Control Subjects. Int J Endocrinol. 2018 Aug 7;2018:5406128. doi: 10.1155/2018/5406128. eCollection 2018. PMID 30158974